CLINICAL TRIAL: NCT00571779
Title: Thoracoscopically-Assisted Epicardial Bilateral Pulmonary Vein Isolations Using the AtriCure Bipolar System and Exclusion of the Left Atrial Appendage for the Treatment of Atrial Fibrillation
Brief Title: AtriCure Minimally Invasive Surgical Ablation for Atrial Fibrillation/RESTORE IIB
Acronym: RESTORE SR IIB
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Other Study IDs: CP2007-2
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

INTERVENTIONS:
Device: AtriCure Bipolar System

SUMMARY:
Feasibility study arm to evaluate the safety of adding the left atrial linear connecting lesions of the Cox-Maze lesion set to the current RESTORE SR II IDE study procedure of performing pulmonary vein isolation, selected left atrial autonomic ganglionated plexi (GP) ablation, and optional left atrial appendage (LAA) excision/exclusion on a beating heart for patients with permanent or persistent Atrial Fibrillation (AF).

ELIGIBILITY:
Inclusion Criteria:

1. Patient between 18 and 80 years of age
2. Patient with documented symptomatic persistent or permanent AF and failure or intolerance of one or more Class I or Class III antiarrhythmic drugs.

   * Persistent AF: AF that is not self-terminating or is terminated electrically or pharmacologically.
   * Longstanding AF: Persistent AF of 12 months (or longer) duration.
   * Permanent AF: Longstanding AF in which electrical or pharmacological cardioversion has failed or has not been attempted.
3. Patient is willing and able to provide written informed consent.
4. Patient has a life expectancy of at least 2 years.
5. Patient is willing and able to attend the scheduled follow-up visits.

Exclusion Criteria:

1. Prior cardiac catheter ablation for the treatment of arrhythmia within 4 months.
2. Patients who refuse, but have not failed and can tolerate anti-arrhythmic medications
3. Myocardial infarction within 8 weeks.
4. Prior cardiac surgery.
5. Patient requires cardiac surgery for treatment other than for AF.
6. Class IV NYHA heart failure symptoms, unless due to uncontrolled AF
7. Cerebrovascular accident within previous 6 months
8. Known carotid artery stenosis greater than 80%
9. Evidence of significant active infection
10. Patient unable to undergo TEE
11. Pregnant woman
12. Patient requires anti-arrhythmic drug therapy for the treatment of ventricular arrhythmia
13. Presence of thrombus in the left atrium
14. Co-morbid condition that in the opinion of the investigator poses undue risk of general anesthesia or port access cardiac surgery
15. Patient is enrolled in another cardiac clinical trial
16. Left ventricular ejection fraction < 30%
17. Left atrial transverse diameter >6.0
18. Patient has undergone previous thoracic targeted radiation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Feasibility of performing the operation by demonstrating the ability to consistently isolate the left and right pulmonary veins and to confirm conduction block across the roof, anterior and LAA linear lesions.
The primary safety endpoint will be determined by assessing the rate of serious adverse events.